CLINICAL TRIAL: NCT03444545
Title: The Performance of a Capnodynamic Method Compared to Transpulmonary Thermodilution in Open Abdominal Surgery
Brief Title: Continous Cardiac Output - Non-Invasive Evaluation (CONNIE)
Acronym: CONNIE
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Anil Gupta, Associate professor in department of pharmacology and physiology, Karolinska Institutet
Other Study IDs: CONNIE 1
Record Dates: First submitted 2018-01-30; First posted 2018-02-23 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Cardiac Output, Low; Cardiac Output, High
Keywords: Cardiac output; Carbon dioxide; Intraoperative monitoring; Pulmonary blood flow
MeSH Terms: conditions — Cardiac Output, Low; Cardiac Output, High

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Capnodynamic method — Expired carbon dioxide is measured with a mainstream infrared sensor (Capnostat-3, Respironics Inc, Wallingford, CT, USA) and gas flow analysed with the flow sensor incorporated in the ventilator (Servo-i, Maquet Critical Care, Solna, Sweden) which was connected to a computer where all the mathematical analysis is carried out with a software written in Matlab™ (The Mathworks Inc, Natick, MA, USA).
  Instead of a fixed ratio between inspiration and expiration, three breaths out of every nine are prolonged with a 3-4 seconds longer expiration creating small changes in end- expiratory CO2
Device: Transpulmonary thermodilution — Each cardiac output measurement comprises an average of three thermodilutions performed successively one after another. TPTD is performed with a PiCCO2 monitor (Pulsion Medical Systems SE, Feldkirchen, Germany)
  Other Names: PiCCO

SUMMARY:
The capnodynamic method non-invasively calculates effective pulmonary blood flow (EPBF) continuously during surgery. In this study EPBF is compared to cardiac output (CO) measured with Transpulmonary Thermodilution (TPTD) att baseline and during hemodynamic changes in patients scheduled for open abdominal surgery at the Karolinska University Hospital, Solna, Sweden.

DETAILED DESCRIPTION:
The capnodynamic method continuously calculates effective pulmonary blood flow (EPBF) with the help of a capnodynamic equation:

ELV x (FACO2(n) - FACO2(n-1)) = deltat(n) x EPBF (CvCO2 - CvCO2(n)) - VTCO2

ELV Effective lung volume [L] EPBF Effective pulmonary blood flow [L/min] n current breath n-1 previous breath FACO2 mean alveolar carbon dioxide fraction CvCO2 mixed venous carbon dioxide content [Lgas/Lblood] CcCO2n pulmonary end-capillary carbon dioxide content [Lgas/Lblood] VTCO2n volume [L] of carbon dioxide eliminated by the current, nth, breath delta t n current breath cycle time [min]

The equation above describes the mole balance between the CO2 delivered to lungs (EPBF), the volume taking part in the gas exchange (ELV) and CO2 excreted from the lungs (VTCO2). Normally there is no difference in CO2 between the actual and the preceding breath as the same amount of CO2 as delivered to the lungs as is excreted. When small changes in CO2 concentration are inserted into the equation obtained with short inspiratory or expiratory pauses in three out of nine breaths, nine different equations are obtained. The three unknown variables; ELV, EPBF and CvCO2can be solved with a linear least square optimization, a well-known numerical mathematical principle. The breathing pattern is automatically controlled by the ventilator which provides continuous calculations of EPBF where each value represents the average of the preceding nine breaths and renews with each breath as the newest replaces the oldest in the equation system.

At the day of surgery, included patients arrive 45 minutes earlier than otherwise at the surgical unit. After safe surgical checklist, vital signs are measured and epidural catheter inserted during a light sedation. Patients are anesthetized and muscle relaxed. An endotracheal tube is inserted in the trachea. Central arterial and vein catheters are inserted in sterile conditions with ultrasound guidance. Anesthesia is maintained with propofol in target controlled infusion and a short acting opioid is added as needed.

The protocol in the first 25 patients comprises simultaneous measurements of EPBF and CO at 1) Baseline (three measurments), 2) PEEP 15cmH2O, 3) PEEP 5cmH2O 4) before epidural activation, 5) 10-15 minutes after epidural activation 6) before volume infusion (when the patient is considered hypovolemic by the attending anaesthesiologist) and 7) shortly after volume infusion.

The attending anesthesiologist has the final responsibility on deciding the order of the protocol, for example if volume infusion should precede PEEP 15 cmH20 if hypovolemia is suspected.

The succeeding 10 patients (patients 26 to 35) are PEEP optimized before start of protocol using a standardiazed open lung tool recruitment. During the PEEP elevation (step 2 in the protocol above) 10cmH2O is added to the optimal PEEP and then released back to the baseline optimal PEEP (step 3).

Each comparative measurement of CO and EPBF in the protocol includes as an average of three TPTD measured with PiCCO2 and and the average of EPBF registered in the beginning of the first TPTD and in the end of the last TPTD.

ELIGIBILITY:
Inclusion Criteria:

* Elective major abdominal surgery requiring advanced hemodynamic monitoring

Exclusion Criteria:

* Symptomatic coronary artery disease, chronic obstructive pulmonary disease with emphysema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having major abdominal surgery requiring advanced hemodynamic monitoring
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Absolute values of EPBF compared to Cardiac output | Mean CO vs EPBF from zero to 4 hours perioperatively
  Mean cardiac output as measured with transpulmonary thermodilution compared to mean effective pulmonary blood flow measured with the capnodynamic method at the start of first thermodilution and during the time interval zero to 4 hours.

SECONDARY OUTCOMES:
Changes in EPBF compared to changes in Cardiac output | Mean CO vs mean EPBF from zero to 4 hours perioperatively
  Measurement of cardiac output and EPBF as described in Outcome 1 before and after hemodynamic changes.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Björne, PhD, Study Director — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sigmundsson TS, Ohman T, Hallback M, Redondo E, Sipmann FS, Wallin M, Oldner A, Hallsjo Sander C, Bjorne H. Performance of a capnodynamic method estimating effective pulmonary blood flow during transient and sustained hypercapnia. J Clin Monit Comput. 2018 Apr;32(2):311-319. doi: 10.1007/s10877-017-0021-3. Epub 2017 May 11. PMID 28497180
- [Background] Sander CH, Sigmundsson T, Hallback M, Sipmann FS, Wallin M, Oldner A, Bjorne H. A modified breathing pattern improves the performance of a continuous capnodynamic method for estimation of effective pulmonary blood flow. J Clin Monit Comput. 2017 Aug;31(4):717-725. doi: 10.1007/s10877-016-9891-z. Epub 2016 Jun 1. PMID 27251701
- [Derived] Sigmundsson TS, Ohman T, Hallback M, Suarez-Sipmann F, Wallin M, Oldner A, Hallsjo-Sander C, Bjorne H. Comparison between capnodynamic and thermodilution method for cardiac output monitoring during major abdominal surgery: An observational study. Eur J Anaesthesiol. 2021 Dec 1;38(12):1242-1252. doi: 10.1097/EJA.0000000000001566. PMID 34155171
- See also: Related Info — http://ki.se/en/fyfa/karolinska-anaesthesia-research-group-for-major-surgery-karisma